CLINICAL TRIAL: NCT02352077
Title: Safety and Efficacy of NeuroRegen Scaffold™ With Bone Marrow Mononuclear Cells or Mesenchymal Stem Cells for Chronic Spinal Cord Injury Repair
Brief Title: NeuroRegen Scaffold™ With Stem Cells for Chronic Spinal Cord Injury Repair
Status: Unknown | Phase: Phase 1 | Type: Interventional
Last Known Status: Enrolling by invitation
Sponsor: Chinese Academy of Sciences (Other Government)
Collaborators: Affiliated Hospital of Logistics University of CAPF (Other); The First Affiliated Hospital of Soochow University (Other); First Hospitals affiliated to the China PLA General Hospital (Other Government)
Responsible Party: Principal Investigator, Jianwu Dai, Principal Investigator of Regenerative Medicine Laboratory, Institute of Genetics and Developmental Biology, CAS, Chinese Academy of Sciences
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAS-XDA-SCI/IGDB
Record Dates: First submitted 2015-01-20; First posted 2015-02-02 (Estimated); Last update posted 2020-12-23 (Actual); Status verified 2016-10

CONDITIONS: Spinal Cord Injury
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- NeuroRegen Scaffold with BMMCs or MSCs transplantation (Experimental)
  Interventions: Biological: NeuroRegen scaffold with BMMCs or MSCs transplantation

INTERVENTIONS:
Biological: NeuroRegen scaffold with BMMCs or MSCs transplantation — Patients with chronic SCI (ASIA grade A) will receive NeuroRegen Scaffold with bone marrow mononuclear cells (BMMCs) or mesenchymal stem cells (MSCs) transplantation after localized scars cleared and after surgery patients will undergo a comprehensive rehabilitation, psychological and nutritional measures.

SUMMARY:
The purpose of this study is to assess the safety and efficacy of NeuroRegen scaffold with bone marrow mononuclear cells (BMMCs) or mesenchymal stem cells (MSCs) in patients with chronic spinal cord injury.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female, 18-65 years old.
2. Completely spinal cord injury at the cervical and thoracic level (C5-T12).
3. Classification ASIA A with no significant further improvement.
4. Patients signed informed consent.
5. Ability and willingness to regular visit to hospital and follow up during the protocol Procedures.

Exclusion Criteria:

1. A current diagnosis of any primary diseases affecting limb functions (e.g., trauma, infection, tumors, congenital malformations, peripheral muscular dystrophy, Huntington's disease, Parkinson's disease).
2. Serious complications (e.g., hydronephrosis due to renal insufficiency, severe bedsores (Ⅲ° above), lower extremity venous thrombosis, severe myositis ossificans).
3. History of life threatening allergic or immune-mediated reaction.
4. Clinically significant abnormalities in routine laboratory examinations (hematology, electrolytes, biochemistry, liver and kidney function tests, urinanalysis).
5. History of mental illness or suicide risk, with a history of epilepsy or other central nervous system disorders.
6. Severe arrhythmias (e.g., ventricular tachycardia, frequent superventricular tachycardia, atrial fibrillation, and atrial flutter) or cardiac degree II or above conduction abnormalities displayed via 12-lead ECG.
7. Lactating and pregnant woman.
8. Alcohol drug abuse /dependence.
9. Participated in any other clinical trials within 3 months before the enrollment.
10. A drug or treatment known to cause effect on the central nervous system during the past four weeks.
11. A drug or treatment known to cause major organ system toxicity during the past four weeks.
12. Poor compliance, difficult to complete the study.
13. Any other conditions that might increase the risk of subjects or interfere with the clinical trial.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Actual)
Dates: Start 2015-01; Primary Completion 2021-12 (Estimated); Study Completion 2021-12 (Estimated)

PRIMARY OUTCOMES:
Safety Evaluation Number of patients with adverse events | 6 months
  Number of patients with adverse events is as a measure of safety and tolerability after collagen scaffold with MSCs transplantation.

SECONDARY OUTCOMES:
Improvements in Neurophysiological Measures omatosensory Evoked Potentials (SSEP) and Motor Evoked Potentials (MEP) monitoring will be assessed | 12 months
  Somatosensory Evoked Potentials (SSEP) and Motor Evoked Potentials (MEP) monitoring will be assessed before and after transplantation.
Improvements in ASIA Impairment Scale | 12 months
  American Spinal Injury Assessment Scale of A, B, C, D or E will be assessed before and after transplantation.
Improvements in Independence Measures and Quality of Life | 12 months
  Functional Independence Measure (FIM) and the Quality of Life Questionnaire (EQ 5D) will be assessed before and after transplantation.
Improvements in Pain assessed based on Visual analog scale (VAS) | 12 months
  Pain intensity will be assessed based on Visual analog scale (VAS) before and after transplantation.
Improvements in Urinary and Bowel Function assessed based on bladder pressure monitory before and after transplantation | 12 months
  The ability to feel and control urination and bowel will be assessed based on bladder pressure monitory before and after transplantation.
Changes at the Transplantation Site in Spinal Cord by Magnetic Resonance Imaging (MRI) | 12 months
  The MRI at the transplantation site will be assessed before and after transplantation.

CONTACTS AND LOCATIONS:
Overall Officials: Jianwu Dai, Ph.D, Principal Investigator — Chinese Academy of Sciences; Sai Zhang, M.D, Study Chair — Affiliated Hospital of Logistics Universtiy of CAPF; Huilin Yang, Ph.D, Study Chair — The First Affiliated Hospital of Soochow University; Shuxun Hou, Study Chair — First Hospitals affiliated to the China PLA General Hospital
Locations (3):
- China (3):
  - First Hospitals affiliated to the China PLA General Hospital, Beijing
  - The First Affiliated Hospital of Soochow University, Suzhou
  - Affiliated Hospital of Logistics Universtiy of CAPF, Tianjin